CLINICAL TRIAL: NCT02521103
Title: A Prospective, Post-market, Multi-center Evaluation of the Clinical Outcomes of the Triathlon TS Total Knee System With Triathlon Tritanium Cone Augments
Brief Title: Triathlon Tritanium Cone Augments Outcomes Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 76
Record Dates: First submitted 2015-07-31; First posted 2015-08-13 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Arthroplasty; Replacement; Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Triathlon Tritanium Cone Augments (Other): Cases who receive the Triathlon TS Total Knee System with at least one Triathlon Tritanium Cone Augment
  Interventions: Device: Triathlon Tritanium Cone Augments

INTERVENTIONS:
Device: Triathlon Tritanium Cone Augments — The Triathlon Tritanium Cone Augments are an extension of the Triathlon Total Stabilizer (TS) system, intended to be used as an optional accessory component in primary or revision TKA

SUMMARY:
This study is a prospective, open-label, post-market, non-randomized, multi-center clinical evaluation of the Triathlon TS Total Knee System with Triathlon Tritanium Cone Augments for revision total knee arthroplasty (TKA) in a consecutive series of patients who meet the eligibility criteria. The revision rate of the Triathlon Tritanium Cone Augments is expected to be less than 2.8% for aseptic loosening of either the Femoral or the Tibial Cone Augments at 2 years postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed an Institutional Review Board (IRB)/Ethics Committee (EC) approved, study specific Informed Patient Consent Form.
* Patient is a male or non-pregnant female, skeletally mature and age 18 years or older at time of study device implantation.
* Patient is a candidate for revision of all femoral and tibial components of a total knee replacement.
* Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

* Patient has a Body Mass Index (BMI) > 45.
* Patient has an active or suspected latent infection in or about the affected knee joint at time of study device implantation.
* Patient has a neuromuscular or neurosensory deficiency, which limits the ability to evaluate the safety and efficacy of the device.
* Patient is diagnosed with a systemic disease (e.g. Lupus Erythematosus) or a metabolic disorder (e.g. Paget's disease) leading to progressive bone deterioration.
* Patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days).
* Patient has a failed unicondylar knee prosthesis.
* Patient has a known sensitivity to device materials.
* Patient is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2015-08; Primary Completion 2025-03-31 (Actual); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of cases with revision of the Femoral Cone Augment or Tibial Cone Augment for aseptic loosening | 2 year

SECONDARY OUTCOMES:
Presence of end-of-stem pain in relation to the Triathlon Tritanium Cone Augments location. | 2 year
  End-of-stem pain is determined via a patient questionnaire; 2 questions are asked in regard to shin and thigh pain location.
Severity of end-of-stem pain. | 2 year
  End-of-stem pain is determined via a patient questionnaire; 2 questions are asked in regard to shin and thigh pain.
  Pain for both the shin and thigh are identified using the following categories:
  * no pain
  * pain with extreme activity only
  * pain with moderate activity
  * pain with normal activity
  * pain at rest
Anderson Orthopaedic Research Institute (AORI) classification and Femoral Cone Augment size. | intraoperative
  The AORI is a bone defect classification which consists of four Types:
  Type I: Metaphyseal bone is intact, with minor bone defects not compromising component stability
  Type IIA: There is metaphyseal bone damage and cancellous bone loss in one femoral/tibial condyle; cement reinforcement, bone grafting or metal augmentation is needed.
  Type IIB: There is metaphyseal bone damage and cancellous bone loss in both femoral/tibial condyles; cement reinforcement, bone grafting or metal augmentation is needed.
  Type III: The metaphyseal bone is deficient and a structural allograft or a custom-made, hinged or revision prosthesis with an extended intramedullary stem is needed
Anderson Orthopaedic Research Institute (AORI) classification and Tibial Symmetric Cone Augment size. | intraoperative
  The AORI is a bone defect classification which consists of four Types:
  Type I: Metaphyseal bone is intact, with minor bone defects not compromising component stability
  Type IIA: There is metaphyseal bone damage and cancellous bone loss in one femoral/tibial condyle; cement reinforcement, bone grafting or metal augmentation is needed.
  Type IIB: There is metaphyseal bone damage and cancellous bone loss in both femoral/tibial condyles; cement reinforcement, bone grafting or metal augmentation is needed.
  Type III: The metaphyseal bone is deficient and a structural allograft or a custom-made, hinged or revision prosthesis with an extended intramedullary stem is needed
Anderson Orthopaedic Research Institute (AORI) classification and Tibial Asymmetric Cone Augment size. | intraoperative
  The AORI is a bone defect classification which consists of four Types:
  Type I: Metaphyseal bone is intact, with minor bone defects not compromising component stability
  Type IIA: There is metaphyseal bone damage and cancellous bone loss in one femoral/tibial condyle; cement reinforcement, bone grafting or metal augmentation is needed.
  Type IIB: There is metaphyseal bone damage and cancellous bone loss in both femoral/tibial condyles; cement reinforcement, bone grafting or metal augmentation is needed.
  Type III: The metaphyseal bone is deficient and a structural allograft or a custom-made, hinged or revision prosthesis with an extended intramedullary stem is needed

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Florida Medical Clinic, Zephyrhills, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Bluegrass Orthopaedics, Lexington, Kentucky
  - The CORE Institute, Novi, Michigan
  - Michigan Heart, St. Joseph Health System, Ypsilanti, Michigan
  - Missouri Orthopaedic Institute, Columbia, Missouri
  - Rothman Institute, Egg Harbor, New Jersey
  - The Orthopaedic Center, Tulsa, Oklahoma
  - Providence Medical Research Center, Spokane, Washington

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT02521103/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT02521103/ICF_001.pdf